CLINICAL TRIAL: NCT05127889
Title: Comparative Evaluation of the Remineralizing Ability of Self-Assembling Peptide P11-4, 2% Arginine Enriched Sodium Fluoride and Functionalized Tri Calcium Phosphate Fluoride Varnishes in Treatment of White Spot Lesions (Randomized Clinical Trial and In Vitro Study)
Brief Title: the Remineralizing Self-Assembling Peptide P11-4, 2% Arginine Enriched Sodium Fluoride and Functionalized Tri Calcium Phosphate Fluoride White Spot Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, bardis Sslah, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED21-3D
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Prevention of White Spot Lesions
Keywords: Wsls,
MeSH Terms: interventions — P11-4 peptide

STUDY DESIGN:
Intervention Model Description: assignment
Who Masked: Participant
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-assembling peptide P11-4 varnish (study group) (Experimental): * Test lesions will be wiped with NaOCl to remove pellicle,
  * Etched for 20 s with 35% H3PO4 Etching Gel to remove mineral deposits on the tooth surface and rinsed with water in accordance with the manufacturer's instructions.
  * The lesions will be dried and isolated with cotton rolls.
  * The varnish will be applied and left undisturbed for 5minutes (till disappearance) to allow diffusion of self-assembly.
  Interventions: Drug: curodont
- Arginine-enriched Sodium Fluoride varnish (study group) (Experimental): * The Arginine powder will be suspended at 2%.
  * A 10 mL of 5% sodium fluoride varnish tube dispensed in a sterile container.
  * 200 mg of Arginine will be vigorously mixed with the varnish matrix for 60 sec using a sterile microbrush.
  * After dryness of the white spot lesion, the prepared varnish will be applied evenly using the micro brush.
  * After application the patient will be instructed to avoid rinsing, eating soft diet and avoid hot drinks for 2 hrs.
  Interventions: Drug: curodont
- Tri Calcium Phosphate Fluoride varnish (positive control group) (Active Comparator): * To limit undesirable oral ingestion, the appropriate dose for the patient will be determined with the help of the dosing guide.
  * The varnish will be mixed with the brush to avoid separation of the material during storage
  * However, to guarantee the best results suction will be used during application of the varnish.
  * A thin uniform layer of the varnish will be applied on the lesion surface by using the supplied brush
  * The applicator brush won't be moved through accumulated saliva to prevent premature setting on the bristles.
  * After application the patient will be instructed to close his mouth, avoid rinsing, eating soft diet and avoid hot drinks for 4 hrs.
  All patients will be encouraged to maintain good oral hygiene through regular brushing.
  Interventions: Drug: curodont

INTERVENTIONS:
Drug: curodont — * To limit undesirable oral ingestion, the appropriate dose for the patient will be determined with the help of the dosing guide.
  * The varnish will be mixed with the brush to avoid separation of the material during storage
  * However, to guarantee the best results suction will be used during application of the varnish.
  * A thin uniform layer of the varnish will be applied on the lesion surface by using the supplied brush
  * The applicator brush won't be moved through accumulated saliva to prevent premature setting on the bristles.
  * After application the patient will be instructed to close his mouth, avoid rinsing, eating soft diet and avoid hot drinks for 4 hrs.

SUMMARY:
The aim of the current study is to compare the remineralizing ability of Self-assembling peptide P11-4, 2% Arginine Enriched Sodium Fluoride and Functionalized Tri Calcium Phosphate Fluoride varnishes in treatment of white spot lesions both in-vivo and in-vitro .

A) Primary Objective

Assessment of:

* Dimensions of the WSLs through digital photography.
* The color of WSLs through spectrophotometer. B) Secondary Objectives

Assessment of:

• Degree of remineralization using Polarized Light Microscope.

DETAILED DESCRIPTION:
White spot lesions (WSLs), defined as "white opacity," occur as a result of subsurface enamel demineralization that is located on smooth surfaces of teeth. The reason of the white appearance is the changes in light-scattering optical properties of the decalcified enamel. The aim of the current study is to compare the remineralizing ability of Self-assembling peptide P11-4, 2% Arginine Enriched Sodium Fluoride and Functionalized Tri Calcium Phosphate Fluoride varnishes

A) Primary Objective

Assessment of:

* Dimensions of the WSLs through digital photography.
* The color of WSLs through spectrophotometer. B) Secondary Objectives

Assessment of:

• Degree of remineralization using Polarized Light Microscope.

PICOTS:

• P - Participants: Children in the age group of 8-12 years having early demineralized carious lesions (WSLs).

* I - Intervention: -Self-assembling peptide P11-4 varnish

  * Arginine enriched Sodium Fluoride varnish C- Comparison:- Functionalized Tri Calcium Phosphate Fluoride varnish
* O -Outcomes:- Reduction in WSLs dimensions and color improvement.

  * Reduction in degree of demineralization of WSLs.
* T- Time: study period will be over 9 months.
* S- Study design: Randomized Controlled Trial (RCT) and in vitro study

This study will consist of two parts: in vivo part (RCT) and in vitro part:

1. In vivo part:

   • Study design: Randomized controlled trial (RCT)

   • Grouping:

   Patients will be randomly allocated into one of the three groups (13/each):

   Group 1: Self-assembling peptide P11-4 varnish (study group) Group 2: Arginine-enriched Sodium Fluoride varnish (study group) Group 3: Tri Calcium Phosphate Fluoride varnish (positive control group)

   Materials used in the study:

   • Self-assembling-peptide (P11-4)
   * Fluoride varnish with TCP5%
   * L-Arginine Sodium Fluoride Varnish
   * Clinical procedures:

   All interventions will be performed by the primary investigator as follows:

   • The dental plaque deposit has to be removed before the assessment. Dental prophylaxis will be performed with a bristle brush and non-fluoridated prophylactic paste during the initial clinical examination and before any examination.
   * photographic assessment by digital camera and color change( E) readings by digital spectrophotometer ( VITA Easy shade) will be performed at 0 , 3 months, 6 months and 9 months throughout the study period for all the patients.
   * During the photographic assessment, all the photographs will be taken with digital camera, Macro lens configuration will be used, the image quality will be set as fine and ISO sensitivity 200. All images will be saved as Joint Photographic Experts Group (JPEG) files suitable for manipulation with the image analysis software.
   * Patient's confidentiality will be respected through the photographic technique.
   * After digital images captured, they will be downloaded and stored as JPEG. Then the images will be analyzed, and compared with baseline images by Abode Photoshop and Auto CAD
   * The enamel color of each WSL will be measured using the spectrophotometer.
   * All measurements will be performed under standardized ambient conditions to ensure accuracy and reproducibility.
   * Three images will be randomly captured for each lesion and analyzed.

   Group 1 (Self assembling peptide P11-4) Prior to application of the test material the following will be done:

   • Test lesions will be wiped with NaOCl to remove pellicle,
   * Etched for 20 s with 35% H3PO4 Etching Gel to remove mineral deposits on the tooth surface and rinsed with water in accordance with the manufacturer's instructions.
   * The lesions will be dried and isolated with cotton rolls.
   * The varnish will be applied and left undisturbed for 5minutes (till disappearance) to allow diffusion of self-assembly.

   Group 2 (Arginine Enriched Sodium fluoride group) Preparation and application of the varnish as following:

   • The Arginine powder will be suspended at 2%.

   • A 10 mL of 5% sodium fluoride varnish tube dispensed in a sterile container.

   • 200 mg of Arginine will be vigorously mixed with the varnish matrix for 60 sec using a sterile microbrush.

   • After dryness of the white spot lesion, the prepared varnish will be applied evenly using the micro brush.

   • After application the patient will be instructed to avoid rinsing, eating soft diet and avoid hot drinks for 2 hrs.

   Group 3 (Tri Calcium Phosphate fluoride) the material will be applied according to the manufacturing instructions as following:
   * To limit undesirable oral ingestion, the appropriate dose for the patient will be determined with the help of the dosing guide.
   * The varnish will be mixed with the brush to avoid separation of the material during storage
   * However, to guarantee the best results suction will be used during application of the varnish.
   * A thin uniform layer of the varnish will be applied on the lesion surface by using the supplied brush
   * The applicator brush won't be moved through accumulated saliva to prevent premature setting on the bristles.
   * After application the patient will be instructed to close his mouth, avoid rinsing, eating soft diet and avoid hot drinks for 4 hrs.

   All patients will be encouraged to maintain good oral hygiene through regular brushing.

   Follow up

   Patients will be recalled for further applications after 3 and 6 months (20) and for WSLs assessment after 3, 6, 9 months.

   Outcome measurement:

   Photographic assessment and color change reading outcomes will be assessed by two other blinded calibrated examiners at the following periods:

1. Baseline 2. 3-month evaluation 3. 6-month evaluation 4. 9-month evaluation

Photographic assessment:

The following will be determined, from photographs for all the patients in relation to WSLs:

1. The area of the labial surface of the tooth
2. WSL area
3. The area of WSL to area of the labial surface of the tooth ratio percent (Percent of WSL)
4. The percentage of WSL ratio related to initial condition at the measured time (Relative Percent)
5. The percentage of decrease in WSL ratio due to time (Percent Decrease)
6. The decrease in the WSL area related to the initial condition (Relative Decrease) Color change readings

   * The values of L* (differences in lightness munsell system ranging from O (black) to 100 (white)), a* (green-red coordinate), and b* (blue yellow coordinate) will be recorded for the WSL and the adjacent sound enamel.
   * Color change, will be calculated as the color difference between the treated and untreated enamel.
   * Participant timeline The study interventions are expected to be conducted from 2021 until 2023.

ELIGIBILITY:
Inclusion criteria

* Patients aged from 8 to 12 years old
* Patients who are medically free from any diseases that would cause enamel defects.
* Patients should have WSLs in labial surface of upper or lower permanent anterior teeth with a score of 1 & 2 according to the ICDAS that don't require operative intervention.

Exclusion criteria

* Patients receiving the following medications will be excluded from the study: tetracyclines, any other medication known to stain teeth, any medication causing dry mouth and/or xerostomia.
* Uncooperative patients
* Mouth breathers

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-04-02 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
dimensional and color assessment | 1. Baseline 2. 3-month evaluation 3. 6-month evaluation 4. 9-month evaluation
  Photographic assessment and color change reading outcomes will be assessed by two other blinded calibrated examiners

SECONDARY OUTCOMES:
Evaluation of the remineralizing ability and degree of remineralization of each agent | 1 month
  Polarized Light Microscopy (PLM) will used for evaluation.

IPD SHARING:
Plan to Share IPD: No